CLINICAL TRIAL: NCT04522024
Title: Concomitant Focal Epicardial Cryoablation During Mei Mini Maze Procedure in Treatment of Lone Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Concomitant Focal Epicardial Cryoablation During Mei Mini Maze Procedure in Treatment of Lone Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiaquan Zhu, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-20-019
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Lone Atrial Fibrillation
Keywords: epicardial cryoablation; epicardial radiofrequency ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mei Mini Maze (Active Comparator): Mei Mini Maze procedure (Unilateral thoracoscopic epicardial ablation by radiofrequency energy from left side)
  Interventions: Procedure: Mei Mini Maze procedure
- Mei Mini Maze plus epicardial cryoablation (Experimental): Epicardial focal cryoablation during Mei Mini Maze procedure
  Interventions: Procedure: Epicardial focal cryoablation

INTERVENTIONS:
Procedure: Epicardial focal cryoablation — Epicardial focal cryoablation on the left atrium around right upper pulmonary vein area
  Arms: Mei Mini Maze plus epicardial cryoablation
Procedure: Mei Mini Maze procedure — Unilateral thoracoscopic epicardial ablation by radiofrequency energy from left side
  Arms: Mei Mini Maze

SUMMARY:
Atrial fibrillation (AF) increases risks of stroke, heart failure and sudden death. Single catheter ablation only has a low success rate due to inadequate transmurality and continuity of the lesion lines. Unilateral thoracoscopic epicardial ablation by radiofrequency energy from left side (Mei Mini Maze procedure, 3M procedure) was applied in our institution in the last 10 years, and gained reasonable results. A more attractive hybrid strategy of epicardial and endocardial ablation was tested to improve the treatment of persistent AF in the investigator's hospital (NCT02968056). Preliminary data from this trial found that insufficient ablation around right upper pulmonary vein area was the key point leading to failure or recurrence. In order to overcome this weakness of the current Mei Mini Maze procedure, concomitant focal epicardial cryoablation performed during the operation may reinforce the lesion lines. The hypothesis of the present study is that additional epicardial cryoablation will improve the success rate compared to Mei Mini Maze procedure alone in the treatment of AF.

This study is a prospective randomized controlled trial within a single institution. Lone AF patients admitted to the cardiovascular surgery department of Shanghai Xinhua Hospital will be screened for enrollment of this study. The study will recruit 150 patients in total. The patients will be randomized allocated into Mei Mini Maze procedure group (3M group) and Concomitant epicardial cryoablation group (3M + Cryoablation group). The 3M group patients only have surgical ablation surgery from left thoracoscope as previously reported, while the 3M + Cryoablation group patients will have additional focal epicardial cryoablation around right upper pulmonary vein area after the Mei Mini Maze procedure is done. The ratio of 3M to 3M + cryoablation group is 1:1, so that each group contains 75 patients. The perioperative data is collected, and the patients will be followed for 6 months. The primary outcome is the maintenance of sinus rhythm at 6 months post operation. The secondary outcomes include off antiarrhythmic drug rate, perioperative complications, major cardiovascular events, stroke, left ventricular systolic function, medical expense, serum brain natriuretic peptide level and quality of life. The aim of this study is to evaluate the efficacy and safety of this novel combined procedure of epicardial radiofrequency and cryoablation.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated atrial fibrillation, without structural heart disease.
2. Failed medical treatment
3. Patient admitted with intent to be treated by surgical ablation

Exclusion Criteria:

1. Previous surgical ablation of atrial fibrillation
2. Concomitant other cardiac diseases which require surgery at the same procedure, such as heart valve disease, congenital heart disease, coronary disease, dilated cardiomyopathy etc.
3. With other forms of severe arrhythmia
4. Ejection fraction of left ventricle less than 30%
5. Anteroposterior diameter of left atrial over 60mm
6. Tumor, active infection, pregnancy.
7. Previous surgeries with left thoracotomy, or expected left pleural adhesion, such as history of tuberculosis infection, pleural effusion, pneumothorax etc.
8. Hyperthyroidism
9. Thrombosis within left atrial appendage
10. General conditions too weak to tolerate the surgeries
11. Patient's circumstance that precludes completion of follow-up and/or obtaining information from the 6 months follow-up
12. Other conditions not appropriate for this study based on the investigators' judgments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Sinus rhythm maintenance rate | At 6 months post operation
  Based on ECG and Holter results after the surgery, any non-sinus rhythm lasting >30 seconds captured on ECG at any time will be considered failure to maintain sinus rhythm

SECONDARY OUTCOMES:
Off any antiarrhythmic drug rate | At 6 months post operation
  Off any antiarrhythmic drug rate
Perioperative complications | Within 1 month after the surgery
  Emergent thoracotomy or exploration for bleeding, renal dysfunction requiring new dialysis treatment, respiratory dysfunction requiring prolonged mechanical ventilation with tracheotomy, new pacemaker implantation, and perioperative death
Major cardiovascular events | Within 6 months post operation
  Death, Nonfatal myocardial infarction, re-admission because of heart disease
Rate of new onset stroke | Within 6 months post operation
  New onset of stroke after the surgery, identified by CT or MRI.
Left ventricular systolic function | At 6 months post operation
  Evaluated by ejection fraction from echocardiogram
Costs of treatment | From surgery to 6 months after the surgery
  There are 3 parts. 1. Cost during the first hospitalization; 2. Cost of all the health care from first discharge to 6 months after the surgery, including seeing clinics, medication, re-hospitalization related to atrial fibrillation/surgical complications/new onset of stroke/other atrial fibrillation related complications. 3. Total cost: the combination of the abovementioned two parts.
Serum NT-proBNP level | At 6 months post operation
  The level of serum NT-proBNP
Quality of life evaluated by short form 36 questionnaire | At 6 months post operation

CONTACTS AND LOCATIONS:
Overall Officials: Yaosheng Wang, MD & Ph.D, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine

REFERENCES:
- [Background] Mei J, Ma N, Ding F, Chen Y, Jiang Z, Hu F, Xiao H. Complete thoracoscopic ablation of the left atrium via the left chest for treatment of lone atrial fibrillation. J Thorac Cardiovasc Surg. 2014 Jan;147(1):242-6. doi: 10.1016/j.jtcvs.2012.10.005. Epub 2012 Nov 2. PMID 23122696
- [Background] Boersma LV, Castella M, van Boven W, Berruezo A, Yilmaz A, Nadal M, Sandoval E, Calvo N, Brugada J, Kelder J, Wijffels M, Mont L. Atrial fibrillation catheter ablation versus surgical ablation treatment (FAST): a 2-center randomized clinical trial. Circulation. 2012 Jan 3;125(1):23-30. doi: 10.1161/CIRCULATIONAHA.111.074047. Epub 2011 Nov 14. PMID 22082673
- [Background] Phan K, Phan S, Thiagalingam A, Medi C, Yan TD. Thoracoscopic surgical ablation versus catheter ablation for atrial fibrillation. Eur J Cardiothorac Surg. 2016 Apr;49(4):1044-51. doi: 10.1093/ejcts/ezv180. Epub 2015 May 23. PMID 26003961
- [Background] van der Heijden CAJ, Vroomen M, Luermans JG, Vos R, Crijns HJGM, Gelsomino S, La Meir M, Pison L, Maesen B. Hybrid versus catheter ablation in patients with persistent and longstanding persistent atrial fibrillation: a systematic review and meta-analysisdagger. Eur J Cardiothorac Surg. 2019 Sep 1;56(3):433-443. doi: 10.1093/ejcts/ezy475. PMID 30698685
- [Background] Cox JL, Churyla A, Malaisrie SC, Pham DT, Kruse J, Kislitsina ON, McCarthy PM. A Hybrid Maze Procedure for Long-Standing Persistent Atrial Fibrillation. Ann Thorac Surg. 2019 Feb;107(2):610-618. doi: 10.1016/j.athoracsur.2018.06.064. Epub 2018 Aug 14. PMID 30118714
- [Background] Milla F, Skubas N, Briggs WM, Girardi LN, Lee LY, Ko W, Tortolani AJ, Krieger KH, Isom OW, Mack CA. Epicardial beating heart cryoablation using a novel argon-based cryoclamp and linear probe. J Thorac Cardiovasc Surg. 2006 Feb;131(2):403-11. doi: 10.1016/j.jtcvs.2005.10.048. Epub 2006 Jan 18. PMID 16434271
- [Background] Wang W, Jiang Z, Lu R, Liu H, Ma N, Cai J, Tang M, Mei J. Effects of Renal Denervation via Renal Artery Adventitial Cryoablation on Atrial Fibrillation and Cardiac Neural Remodeling. Cardiol Res Pract. 2018 Dec 11;2018:2603025. doi: 10.1155/2018/2603025. eCollection 2018. PMID 30647968
- [Background] Blomstrom-Lundqvist C, Johansson B, Berglin E, Nilsson L, Jensen SM, Thelin S, Holmgren A, Edvardsson N, Kallner G, Blomstrom P. A randomized double-blind study of epicardial left atrial cryoablation for permanent atrial fibrillation in patients undergoing mitral valve surgery: the SWEDish Multicentre Atrial Fibrillation study (SWEDMAF). Eur Heart J. 2007 Dec;28(23):2902-8. doi: 10.1093/eurheartj/ehm378. Epub 2007 Nov 5. PMID 17984136